CLINICAL TRIAL: NCT01414218
Title: Influence of Humor as a Way of Life on Well Being, Quality of Life and Immune Function
Brief Title: The Impact of a Humor Seminar on General Well Being, Quality of Life and Psychological Distress Among Community Dwelling Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Happy Nation Society (Other)
Responsible Party: Freda DeKeyser Ganz, Happy Nation Society
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: humor1
Record Dates: First submitted 2011-08-04; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Improve Mental Health
Keywords: elderly; humor; general well being; psychological distress; health quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Humor as Way of Life Seminar (Experimental): See description of study in previous section for further details.
  Interventions: Behavioral: Humor as a Way of Life Seminar

INTERVENTIONS:
Behavioral: Humor as a Way of Life Seminar — One session per week lasting 2-3 hours per session for 4 months. Sessions will include the videotaping of humorous stories or situations and instruction related to strategies to incorporate humor into everyday life.

SUMMARY:
1. Senior citizens living in the community who participate in a humor seminar will have improved health quality of life compared to those not participating in the seminar.
2. Senior citizens living in the community who participate in a humor seminar will have improved general well being compared to those not participating in the seminar
3. Senior citizens living in the community who participate in a humor seminar will have decreased psychological distress compared to those not participating in the seminar

DETAILED DESCRIPTION:
Participants for this study will be chosen from senior centers . All members of the senior centers who can read and write either Hebrew or English and are not cognitively impaired (as assessed by the administrator/social worker in charge of the center) will be asked to participate. It is estimated that between 30-50 members of each senior center will agree to participate. The control group will be chosen by convenience sampling of members from other, different senior centers. These centers will be chosen based on close geographic proximity and similar demographic characteristics to the experimental, humor group, senior centers. The choice of which center will be used for the experimental and control groups will be based on logistic considerations.

This method of sample selection and group assignment were chosen due to several considerations. At present there are approximately 60 participants in the Rishon Lezion Holocaust survivor senior center. It is highly unlikely that all of the members of the center will agree to participate in the study and/or will continue with the entire intervention. Based on a power of .80 and an alpha rate of .05, in order to detect a significant difference between two groups with a moderate effect size, a total of 64 subjects will be necessary for each of the two groups, the experimental and the control each group. Therefore, there are not enough seniors in one center to participate in either groups and additional sites for subject recruitment was found to be necessary.

A second consideration is diffusion of the treatment protocol. It is thought that if both the control and humor groups were recruited from the same senior center, then there would be the possibility that the seniors would discuss among themselves the humor intervention, thereby leading to a diffusion of treatment. In this situation, it might be hard to differentiate between those who participated in the humor and the control group. Therefore, the seniors of the control group would need to be recruited from another senior center.

This process then leads to another issue, namely selection bias, in that the control and humor groups might be different from the outset of the study. Two measures will be taken to decrease this threat to the internal validity of the study. Firstly, an attempt will be made to match the senior centers that will be used to recruit those in the control group with the senior centers used for the humor group, based on geographic location and demographic characteristics. Secondly, both the control and humor groups will be asked to complete the questionnaires at the beginning and at the end of the study. Therefore, differences will be determined between the two groups at two points in time.

Humor Program: The "Humor as a Way of Life" program will be comprised of one session per week lasting 2-3 hours per session. The program will take six months to complete. The first three months of the program will be moderated by Mr. Yochanan Waller, a known video producer and humorist. Under Mr Waller's direction, each participant will be requested to relate a humorous story or situation. These sessions will be video recorded. Between each session, Mr Waller will edit each session. At the next session, all of the participants will view all of the stories related during the previous session. Any parts of the videos that are not used for the purpose of the program will be destroyed.

The first four weeks of the program will include strategies to incorporate humor into everyday life. These sessions will be conducted by Mr. Enzo Agada, a known humorist, and his wife, Amalia Garbulsky, a Social Worker. The topic of humor and its impact on everyday life will be presented and discussed. Initially the moderator will tell humorous stories and aim to trigger reactions or comments from the participants about their own personal associations of what they just heard. Participants will be asked about humorous life events and will be asked to share those events with the group. During each session the moderators will generate an atmosphere of mirth and will try to involve as many participants as possible in the discussion. The moderator will act as a stimulant for humor, smiling, and laughter.

At the end of the four months, a large celebration will be conducted where a final video will be shown that summarizes the project.

During the next two months, volunteers will be recruited to transport the participants to other senior centers in groups of 3-4. The participants will share with the seniors the final video and will try and encourage other seniors to use humor in their daily lives.

Instruments: Four questionnaires will be used in this study; a demographic data questionnaire, the RAND Health Survey (Hays, Sherbourne, & Mazel, 1993), the General Well Being Schedule (Dupuy, 1987)and the Brief Symptom Inventory (Derogatis & Spencer, 1982).

After institutional ethical review and approval, each potential senior center administrator will be contacted to gain approval for admission to the site to collect data. The principle investigator of the study will oversee and supervise all data collection. All members of each senior center who speak and write Hebrew or English and are cognitively competent (as assessed by the administrator/social worker of each senior center) will be asked to participate. These seniors will be contacted, the study will be described and informed consent obtained. Copies of the informed consent form will be given to each participant. After informed consent was obtained, each participant will fill out the three questionnaires. Data collectors will be available to help participants fill out their forms if necessary. This data collection will take place before the project has begun. Each participant will be asked to write the last four digits of their identity numbers on the form so that follow up questionnaires will be able to be correlated with baseline data. All subjects will fill out all forms at baseline and after six months, after completion of the project. Control subjects will be offered the option of participating in the next humor therapy session whenever possible.

If the results of the GWB questionnaire indicate great psychological distress of the participant, then the administrator/social worker of the senior center will be informed as necessary.

Analysis: Descriptive statistics will be used to describe the sample and results of the RAND and GWB questionnaires. Differences between the two groups will be determined using a MANOVA.

ELIGIBILITY:
Inclusion Criteria:

* attendance at a community senior center
* ability to read and write hebrew or English

Exclusion Criteria:

* Not cognitively impaired

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
General Well Being | after 6 months
  General Well Being as measured by the General Well Being Scale
Psychological Distress | after 6 months
  Psychological distress as measured by the Brief Symptom Inventory
Health Quality of Life | after 6 months
  Health Quality of Life as measured by the Rand Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Freda Dekeyser Ganz, PhD, Principal Investigator — Hadassah Hebrew University